CLINICAL TRIAL: NCT01407939
Title: Efficacy of Bitter Taste Blockers on Flavor Acceptance in Pediatric Populations
Brief Title: Efficacy of Bitter Blockers on Taste Perception in Children and Adults
Acronym: BL
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Julie A. Mennella, Member, Monell Chemical Senses Center
Other Study IDs: 809789; 1R01DC011287-01 (NIH)
Record Dates: First submitted 2011-07-19; First posted 2011-08-02 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Healthy
Keywords: Bitter Taste; Bitter Blockers; Pediatric Medications; Sensory methodology; Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Children, Adults: 3- to 15-year old children and their parent (adults

SUMMARY:
This proposal describes 2 basic research studies that will be conducted sequentially. Study 1 will test the efficacy of both classic and newly developed "generally recognized as a safe" (GRAS) bitter blockers on the perceived bitterness and acceptance of different classes of bitter-tasting compounds by children and compare their responses to adults. Because variations among and between children and adults in terms of sensitivity to different bitter compounds are due in part to genetically determined receptor variation, the investigators will consider genotype when assessing how well bitter blockers perform. In Study 2, the investigators aim to evaluate different methods (forced-choice procedures, hedonic face scales) used for testing children to determine their reliability and reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, term children of either sex and all races/ethnicities will be eligible for this study.
* Children must be between 3 and 10 years of age.

Exclusion Criteria:

* Children who are on any medications that may alter taste sensitivity
* Mothers who are pregnant

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Total number of subjects to be enrolled into the study: 300 mothers and 300 children (ages 3-10) =600 total subjects.
  Mothers will be recruited from the community of greater Philadelphia through newspaper and online ads and initial interviews are conducted over the telephone.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2011-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who rate bitter solutions with added bitter blockers as less bitter than the bitter solution alone. | 2 hours
  Primary outcome variables are the proportion of subjects by age group (children and adults) judging a variety of GRAS bitter compounds with a bitter blocker as less bitter or more pleasant than the bitter compound alone (the efficacy of the bitter blocker). At least 5 bitter compounds and 5 GRAS bitter blockers will be used. We will determine how these measures are affected by the age and genotype of the subjects.

SECONDARY OUTCOMES:
Biometrics and Genotype | One year
  For both Studies 1 and 2, the secondary outcome variables include age, genotype of various taste receptor genes (e.g., TAS2R38, TAS2R20, TAS2R31), body weight and height.
Differences in bitterness ratings obtained via different pediatric taste-assessment methodologies. | 2 hours
  We will determine whether the bitter-blocker pairings assessed as most effective by the children using the forced-comparison procedure (bitter alone vs bitter plus blocker) yield statistically different ratings when children use a 3-point, 5-point, or 7-point scale (with happy and sad faces to denote the degree of liking and disliking) after children, of varying ages, taste each of these solutions.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Mennella, PhD, Principal Investigator — Monell Chemical Senses Center
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Mennella JA, Roberts KM, Mathew PS, Reed DR. Children's perceptions about medicines: individual differences and taste. BMC Pediatr. 2015 Sep 21;15:130. doi: 10.1186/s12887-015-0447-z. PMID 26391354
- [Derived] Mennella JA, Reed DR, Roberts KM, Mathew PS, Mansfield CJ. Age-related differences in bitter taste and efficacy of bitter blockers. PLoS One. 2014 Jul 22;9(7):e103107. doi: 10.1371/journal.pone.0103107. eCollection 2014. PMID 25050705